CLINICAL TRIAL: NCT00587249
Title: Phase I Trial of ICC-1132, a Candidate Vaccine Against Plasmodium Falciparum Malaria Based on a Viral-like Particle Comprising Recombinant Hepatitis B Core Antigen and Circumsporozoite Epitopes, to Assess Vaccine Safety and Immunogenicity in Healthy Adult Volunteers
Brief Title: ICC-1132 - Candidate Vaccine Against P Falciparum Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-416; CVD 16000
Record Dates: First submitted 2008-01-03; First posted 2008-01-07 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-03

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria, Plasmodium falciparium, Hepatitis B Core Antigen, Circumsporozoite Epitopes
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Aluminum Hydroxide

ARMS (3):
- 3 (Experimental): 50 mcg of ICC-1132 with alhydrogel adjuvant.
  Interventions: Biological: Malaria ICC-1132; Biological: Alhydrogel
- 2 (Experimental): 20 mcg of ICC-1132 with alhydrogel adjuvant.
  Interventions: Biological: Malaria ICC-1132; Biological: Alhydrogel
- 1 (Experimental): 10 mcg of ICC-1132 with alhydrogel adjuvant.
  Interventions: Biological: Malaria ICC-1132; Biological: Alhydrogel

INTERVENTIONS:
Biological: Malaria ICC-1132 — ICC-1132, a candidate malaria vaccine, with alhydrogel will be in 2 ml glass vials containing ICC-1132 at either 40 mcg/ml or 100 mcg/ml concentration formulated with alhydrogel at 1mg/ml. Each vial will contain approximately 0.8 ml solution to permit recovery of 0.5 ml for injection. When shaken, the solution is off-white to greyish-white turbid liquid free of foreign particulate matter.
Biological: Alhydrogel — Aluminum hydroxide gel.

SUMMARY:
The purposes of this study are to evaluate the safety and immune responses (the body's defense system) to an investigational malaria vaccine called ICC-1132. Three different doses of the vaccine will be studied in 3 groups of people, and the results will be compared. The study will involve about 80 healthy volunteers, 18-45 years of age, who will receive an injection of a specific dose of the vaccine in their arm on 2 or 3 different days. Blood samples will be collected approximately 15 times for laboratory studies. Volunteers will record their temperature twice per day. Volunteers will complete a daily symptom diary for 7 days after each vaccination. Volunteers will participate in the study for up to 13 months.

DETAILED DESCRIPTION:
This is a Phase I, dose-escalating clinical trial of a candidate malaria vaccine, ICC-1132. The primary objective is to assess and compare the safety, reactogenicity, and immunogenicity of 3 intramuscular injections of ICC-1132. The vaccine is absorbed to alhydrogel adjuvant. Three dose levels, 10 mcg, 20 mcg, and 50 mcg, will be compared. Vaccine will be injected intramuscularly on study days 0, 56 +/- 4 and 168 +/- 14, with the exception of the 10 mcg dose cohort which will receive only 2 injections, 1 each at 0 and 2 months. The study was originally designed as a blinded, dose-escalating trial comparing 3 doses (10, 20, and 50 mcg) of ICC-1132 in saline to 3 doses of ICC-1132 + alhydrogel (10, 20, and 50 mcg). Prior to removing the saline formulated ICC-1132 from the trial, the first 16 eligible volunteers were assigned to the 10 mcg cohort, with 8 receiving ICC-1132 in saline and 8 receiving ICC-1132 + alhydrogel. The next 3 eligible volunteers were assigned to the 20 mcg cohort and were randomly assigned to receive ICC-1132 in saline or ICC-1132 + alhydrogel. The study will continue with vaccinations using only the alhydrogel formulation of the vaccine. Subjects will be observed for immediate localized or systemic reactions for 30 minutes before being released from the clinic. Vital signs and a post-vaccination arm check will be performed approximately 30 minutes after vaccine administration. Subjects will return to the outpatient clinic for clinical examinations at 24 +/- 6 and 48 +/- 6 hours, and at days 7 +/- 1, 14 +/- 2, and 28 +/- 4 after each vaccination. Volunteers will complete a daily symptom diary for 7 days after each vaccination. Additional follow up visits will be done 84 +/- 7 days after the second vaccine and 56 +/- 7 days after the third vaccine. A telephone interview will be done at day 4 +/- 1 after each immunization and 168 +/- 14 days after the third immunization. Participants will be involved in study related procedures for up to 393 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 45 years of age.
* Willingness to participate in this study as evidenced by a signed, written informed consent.
* An informed consent written exam score of at least 70%.
* If female, willingness to avoid pregnancy and practice adequate birth control from the time of study enrollment until at least 2 months after the third vaccination.
* Agrees to refrain from blood donation during the course of the study.
* Agrees to be available for all scheduled study visits (vaccinations and follow-up).
* Agrees not to participate in concurrent vaccine or drug trials other than those evaluating Apovia's ICC-1132.

Exclusion Criteria:

-Evidence of renal disease, as indicated by any of the following: Creatinine >1.5 mg/dL within the 7 days before first vaccination RBC or WBC casts in urine Urine protein greater than or equal to 1 plus on urinalysis

-Evidence of cardiovascular disease, as indicated by any of the following: BP >150/90 mmHg in two measurements on different days Hospitalization for heart attack, arrhythmia, or syncope Murmur (other than a functional murmur) detected on physical examination

* History of cancer (except basal call carcinoma of the skin and cervical carcinoma in situ)
* Evidence of liver or other reticuloendothelial disease, as indicated by any of the following:

Positive serology for hepatitis B surface antigen Positive serology for hepatitis C antibody AST or ALT more than 1.5 times normal within the 7 days before first vaccination Hepatosplenomegaly, jaundice, or lymphadenopathy on physical examination

-Evidence of neurological disease, as indicated by any of the following: History of seizures (other than febrile seizures as a child <5 years old) History of unconsciousness (other than a single brief "concussion") Recurrent severe headaches or a diagnosis of migraine headaches Focal neurological deficit on physical examination suggesting a pathologic process

-Evidence of gastrointestinal disease, as indicated by any of the following: Recurrent diarrhea (>5 episodes during the past 6 months, each lasting at least 3 days, with at least one week between episodes) Frequent indigestion or heartburn that requires daily antacids or other medical therapy Diagnosed by a doctor as having uncontrolled irritable bowel syndrome, Crohn's disease, ulcerative colitis, celiac disease, or stomach or intestinal ulcers Blood in the stool during the past year (other than occasional small amount from straining or hemorrhoids)

-Evidence of hematologic, rheumatologic, or immunologic disease, as indicated by any of the following: WBC <3.0 x 10^3/mm^3 or >13.5 x 10^3/ mm^3 within the 7 days before first vaccination Absolute neutraophil count <1500/ mm^3 within the 7 days before first vaccination Hemoglobin (within the 7 days before first vaccination)

* Females <10.5 g/dL or >18 g/dL
* Males <11.5 g/dL or >20 g/dL History of greater than or equal to 2 hospitalizations for invasive bacterial infections (pneumonia, meningitis) History of hemoglobinopathy such as sickle cell disease or thalassemia Diagnosis of collagen vascular disease such as lupus or dermatomyositis Positive serology for HIV antibody
* History of diabetes mellitus or a 3-hour fasting blood glucose >125 mg/dL
* Evidence of pulmonary disease as indicated by any of the following:

History of asthma requiring the use of oral medications or metered dose inhalers in the previous 12 months Wheezes, rales, or prolonged expiratory phase on auscultation of the lungs

* Is required to take a daily medication other than vitamins, levothyroxine, birth control pills, hormone replacement therapy for menopause, or the following medications for attention deficit hyperactivity disorder (pemoline [Cylert], methylphenidate HC1 [Ritalin, Ritalin-SR, Concerta], dextroamphetamine sulfate [Dexedrine, Adderall], bupropion HC1 [Wellbutrin, Wellbutrin-SR])
* Receives allergy shots or uses allergy medications chronically
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Pregnancy (positive urine pregnancy test immediately prior to each dose, or positive serum pregnancy test during screening) or breastfeeding
* Temperature >38 degrees C (100.4 degrees F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis on vaccination day; subjects may be rescheduled to enter the trial after illness has resolved, as per protocol
* Use of investigational drugs, products or devices within 30 days prior to study drug administration
* Vaccination with live vaccine within 30 days or killed vaccine within 2 weeks
* History of malaria infection or vaccination with candidate malaria vaccine
* Allergy to aminoglycosides, tetracycline, or related antibiotics such as gentamicin, kanamycin or doxycycline
* Weight less than 110 pounds
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol
* History of immediate-type hypersensitivity reaction to any vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2002-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Provide a preliminary assessment of the safety of ICC-1132 plus alhydrogel in healthy adults and to determine if there are any probable or definitive SAEs. | Duration of study.

SECONDARY OUTCOMES:
Immunogenicity of ICC-1132 plus alhydrogel in healthy human subjects. | Serum will be collected at the time of each immunization and at 14 and 28 days after each immunization. Day 84 following the 2nd immunization and at Day 56 after the 3rd vaccination and possibly at Day 168 after the 3rd vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Gregson AL, Oliveira G, Othoro C, Calvo-Calle JM, Thorton GB, Nardin E, Edelman R. Phase I trial of an alhydrogel adjuvanted hepatitis B core virus-like particle containing epitopes of Plasmodium falciparum circumsporozoite protein. PLoS One. 2008 Feb 6;3(2):e1556. doi: 10.1371/journal.pone.0001556. PMID 18253503